CLINICAL TRIAL: NCT01318590
Title: Prospective Study on Endoscopic Ultrasound (EUS) Celiac Bloc Efficacy in Chronic Pancreatitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Closed by CHUM REB for incomplete documentation of research activities.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); Erasme University Hospital (Other)
Responsible Party: Principal Investigator, A Sahai, Gastroenterologist, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CE 10 160
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Pancreatitis, Chronic
Keywords: Pancreatitis, Chronic; Abdominal Pain; Celiac bloc; Endosonography
MeSH Terms: conditions — Pancreatitis, Chronic; Abdominal Pain | interventions — Pharmaceutical Preparations; Bupivacaine; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Celiac bloc (Experimental): The experimental arm will consist of the fractional injection on both sides of the celiac trunk, via EUS, of a local anesthetic (10 ml of Bupivacaine 0.5% (gr / ml)) and an injection of steroids (Triamcinolone 40 mg). In this group antibiotic prophylaxis will be administered after administration of sedation (Cephazolin 1gr IV or Gentamycin).
  Interventions: Drug: EUS procedure with drug injection
- Conservative treatment (Sham Comparator): Subject will undergo standard EUS without any additional interventions.
  Interventions: Other: EUS procedure

INTERVENTIONS:
Drug: EUS procedure with drug injection — EUS procedure with injection of 10 ml Bupivacaine 0.5% and 40 mg of Triamcinolone in the celiac plexus after administration of intravenous (IV) antibioprophylaxis
  Other Names: Bupivacaine & Triamcinolone Acetonide injection in the celiac plexus
  Arms: Celiac bloc
Other: EUS procedure — EUS procedure without any drug injection
  Arms: Conservative treatment

SUMMARY:
The purpose of this study is to determine if celiac bloc (with injection of steroid and local anesthetic) is superior to a sham procedure for pain control and quality of life improvement in patient with chronic pancreatitis and abdominal pain.

DETAILED DESCRIPTION:
Chronic pancreatitis is a condition that can lead to very disabling pain symptoms that are difficult to control. The use of morphine is often necessary and also induces a series of secondary symptoms.

In this context, the injection into the celiac plexus block of a local anesthetic has often been proposed as an alternative. This procedure, by interrupting the afferent pain signal of pancreatic origin, aims to reduce pain and improve quality of life at the cost of fewer side effects.

This procedure can be performed transcutaneously using the anatomical landmark or under radiological control. It can also be performed via endosonography (EUS) with better control of the injection site under ultrasound control.

The results of the literature concerning the efficacy of the celiac block in chronic pancreatitis are rather encouraging with reported figures of partial or complete pain control in 39 to 65% of patients [1-7].

However, the number of prospective studies concerning this technique performed endoscopically remains low to date. In particular, there are no case control studies. Data is also poor on the impact on quality of life.

The study proposed here will therefore attempt to provide answers to the questions still pending: is the block by EUS superior to a diagnostic EUS without treatment? ; how long does this treatment last? ; does it have an impact on the quality of life of patients? This study and its draft are inspired by a similar recent study conducted in our department on patients with pancreatic neoplasia. The results of the latter are being submitted for publication.

ELIGIBILITY:
Inclusion Criteria:

* abdominal pain compatible with pancreatic ethiology since at least 3 months
* chronic pancreatitis on Computed Tomography (CT), Endoscopic Retrograde Cholangiopancreatography (ERCP) or EUS
* EUS feasible
* inform consent

Exclusion Criteria:

* pregnant women
* allergy to local anesthetic
* acute pancreatitis in the last 2 weeks
* suspicious lesion on pancreatic EUS examination
* celiac bloc in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-11-18 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Pain reduction on Likert scale | each month for six months
  Pain scale with 7 levels

SECONDARY OUTCOMES:
Quality of Life (QOL) score | each month for six months
  the digestive disease QOL questionnaire 15 (DDQ-15) is used to analyze QOL

CONTACTS AND LOCATIONS:
Overall Officials: Anand V Sahai, MD, Principal Investigator — CHUM
Locations (2):
- Erasme Hospital, Brussels, Belgium
- CHUM, Montreal, Quebec, Canada